CLINICAL TRIAL: NCT07005947
Title: Long COVID-19 Cutaneous Signatures: An ARPA Funded Research Project
Acronym: LCCS
Status: Recruiting | Type: Observational
Sponsor: CND Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: The LCCS Study
Record Dates: First submitted 2025-06-03; First posted 2025-06-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Long COVID-19; Acute COVID-19; Postural Orthostatic Tachycardia Syndrome (POTS); Diabetic Neuropathy
Keywords: COVID; Diabetic Neuropathy; Postural orthostatic tachycardia syndrome; POTS
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Three skin biopsies and one plasma blood collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Long COVID: Participants with Long COVID
- Acute COVID: Participants with acute COVID who tested positive for COVID without persistent symptoms
- Postural Orthostatic Tachycardia Syndrome (POTS): Participants with postural orthostatic tachycardia syndrome (POTS)
- Diabetic neuropathy: Participants with diabetic neuropathy

SUMMARY:
This is a prospective, longitudinal study involving 300 participants for a single visit to compare Long COVID-19 neurocutaneous biosignatures with those of other disorders affecting the sensory and autonomic nervous system.

DETAILED DESCRIPTION:
This is a prospective, longitudinal study involving 300 participants for a single visit to compare Long COVID-19 neurocutaneous biosignatures with those of other disorders affecting the sensory and autonomic nervous system. The evaluations will include clinical assessments, neurologic exams, patient reported outcome surveys, and skin biopsies from three locations. Data will be collected on the amount of P-SYN in cutaneous nerve fibers. The cohorts of interest are as follows:

1. 100 participants with Long COVID-19 defined by NIH PASC criteria
2. 100 participants with acute COVID-19 who tested positive for COVID-19 without persistent symptoms defined WHO criteria
3. 50 participants with postural orthostatic tachycardia syndrome (POTS)
4. 50 participants with diabetic neuropathy

There are no plans for additional visits at this time.

If interested to learn more about this study, please complete the form here for someone to contact you. "here" would take you to the said form.

ELIGIBILITY:
Inclusion Criteria, just one of the following:

* Long COVID-19 defined by NIH PASC criteria OR
* Acute COVID-19 who tested positive for COVID-19 without persistent symptoms OR
* Postural orthostatic tachycardia syndrome (POTS) OR
* Diabetic neuropathy

Exclusion Criteria:

* Clinical evidence of severe peripheral vascular disease
* History of ulceration, poor wound healing or vascular claudication
* History of allergic reaction to local anesthesia (for biopsy collection)
* Use of oral anticoagulants (aspirin or Plavix alone is allowed)
* History of a bleeding disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and females ages 18-80 who have been diagnosed with one of the following:
  1. Long COVID defined by NIH PASC criteria OR 2. Acute COVID who tested positive for COVID without persistent symptoms OR 3. Postural orthostatic tachycardia syndrome (POTS) OR 4. Diabetic neuropathy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-16 (Estimated)

PRIMARY OUTCOMES:
Pathology and nervous system changes that occur in patients suffering from sensory and autonomic function changes | Current - December 31,2025
  This is a single site study of subjects with Long COVID, subject with a previous positive COVID test without persistent symptoms, and POTS subjects and diabetics. Neurocutaneous biosignatures will provide insight into the pathology and nervous system changes that occur in patients suffering from sensory and autonomic function changes.

CONTACTS AND LOCATIONS:
Locations (1):
- CND Life Sciences, Scottsdale, Arizona, United States